CLINICAL TRIAL: NCT03342482
Title: Glutamate Neuro-Excitotoxicity in GWI
Acronym: GWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University (Other)
Collaborators: Georgetown University (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kathleen Holton, Assistant Professor, American University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-2017-301
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Gulf War Syndrome
Keywords: MSG; Gulf War Syndrome; Diet; Glutamate
MeSH Terms: conditions — Persian Gulf Syndrome

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to immediately start a one-month dietary intervention restricting consumption of glutamate, or will be waitlisted as a control group for the first month, and then will begin the one-month dietary intervention period (which will be completed at home). Then subjects will return to DC, will complete all measures again, and then will participate in a double-blind, placebo-controlled, crossover challenge with MSG and placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 5 g of placebo (sugar and salt) will be administered in veggie capsules
  Interventions: Other: Low-glutamate diet
- MSG (Experimental): 5 grams of MSG will be administered in veggie capsules
  Interventions: Other: Low-glutamate diet

INTERVENTIONS:
Other: Low-glutamate diet — The dietary intervention consists of a one-month low-glutamate diet, followed by a randomized crossover challenge with MSG and placebo to measure return of symptoms.

SUMMARY:
The objective of the proposed research is to examine whether dietary exposure to food additives containing glutamate may be contributing to symptoms in Gulf War Illness (GWI). The rationale for proposed study comes from data in the fibromyalgia field which suggests that reducing the consumption of dietary glutamate can reduce over-excitation in the nervous system, leading to symptom improvement. In prior research, a low-glutamate diet (restricting food additive consumption) was tested in fibromyalgia patients. After one-month on the diet, 84% of patients had >30% of their symptoms go away (with 11 symptoms remitting on average), and 8 subjects had complete remission of all symptoms. Subjects then had a significant return of symptoms upon challenge with monosodium glutamate (MSG) as compared to placebo. Since there is almost complete symptom overlap between fibromyalgia and GWI, it is of utmost importance to test this diet as a low-cost treatment option in GWI patients.

The findings from this research will ultimately be applicable to all GWI patients and potentially to other veterans with a similar symptom profile as well. The ultimate impact of this research could be quite profound, as it has the potential to impact all of the symptoms of GWI, as opposed to being a proposed treatment for only one of the symptoms. This dietary treatment has been shown to dramatically affect symptoms like fatigue, cognitive dysfunction, and pain; and thus, has the potential to dramatically improve quality of life for these individuals. Potential benefits of the treatment are great, and risks are minimal, as the treatment involves shifting the diet to a healthier, whole-food approach.

First, the study will confirm or negate the idea that abnormal glutamate signaling in the nervous system could be causing symptoms in GWI. Second, if found to be successful, then this will provide a low-cost, easy-to-implement treatment option for the many veterans suffering from this multi-symptom illness. Third, this research could lead to future studies to identify potential causes of this abnormal neurotransmission, to help prevent future illness onset.

DETAILED DESCRIPTION:
Objective/ Hypothesis: The objective of this clinical trial is to test the effectiveness of a low-glutamate diet in GWI patients, as a way to mediate symptom occurrence by reducing excess glutamatergic neurotransmission.

Specific Aims:

Aim 1- Determine if GWI is a glutamate neurotoxicity disorder, by testing whether reduced exposure to dietary glutamate can modulate symptoms. Hypothesis: Dietary glutamate restriction will significantly reduce GWI symptoms, including fatigue, cognitive dysfunction, pain, problems sleeping, headache/migraine, and diarrhea; as measured by symptom questionnaire, dolorimetery, computerized cognitive testing, EEG and fMRI memory testing. Additionally, brain glutamate levels will be reduced after one month on the diet, as measured by magnetic resonance spectroscopy (MRS).

Aim 2- Confirm that altered dietary glutamate exposure was the cause of symptom improvement.

Hypothesis: Challenge with MSG, as compared to placebo, in a randomized, double-blind, placebo-controlled crossover challenge, will significantly increase the occurrence of symptoms, cause increased pain sensitivity as measured by dolorimetry, increased excitatory neurotransmission as measured by EEG, and a worsening of cognitive function as measured by computerized cognitive testing.

Study Design: 40 subjects will be recruited from around the US . After phone screening, eligible individuals will travel to Washington DC for their first visit, where subjects will undergo baseline testing, including assessment of symptoms, cognition, brain glutamate levels and working memory testing using fMRI. For phase 1, subjects will be randomized to a low-glutamate diet (n=20) or a waitlisted group (n=20 as controls), and symptom occurrence will be compared after one month. Waitlisted participants will follow the low-glutamate diet over the following month. At the end of phase 1, subjects will return to DC, will undergo post-diet assessment of symptoms (same as baseline), and then will move onto Phase 2 of the study, a randomized, double-blind, placebo-controlled crossover challenge, to test whether symptoms recur upon challenge with MSG and not with placebo. Subjects will be randomized as to which contingency (MSG or placebo) is received first, and will receive MSG for 3 consecutive days on one of the weeks and placebo for 3 consecutive days on the other week. Symptoms, EEG and cognition will be assessed on day 3 of challenges each week. All subjects will still be following the low-glutamate diet during the challenge period, so their only exposure to glutamate will be from the week they receive the MSG.

ELIGIBILITY:
Inclusion Criteria:

* Males & Females
* Served (and was deployed) in the Persian Gulf War
* Fulfill both Kansas and CDC definitions of GWI
* Stable medication regimen for 3 or more months

Exclusion Criteria:

* Active Duty Military
* Current substance use disorder
* Unwilling to change diet for 2 months
* Severe asthma requiring past hospitalization
* Seizure disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2020-07-07 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Symptom Score Change | Baseline, 1 month, 5th week, 6th week
  The number and type of symptoms will be assessed with a symptom score measure

SECONDARY OUTCOMES:
Cognitive Function | Baseline, 1 month, 5th week, 6th week
  A computerized cognitive battery will measure cognitive function

OTHER OUTCOMES:
Change in EEG | Baseline, 1 month, 5th week, 6th week
  Electroencephalography will be used to measure brain excitation
Change in Brain Glutamate Levels | Baseline, 1-month
  Brain glutamate levels will be measured using magnetic resonsnance psectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen F Holton, PhD, Principal Investigator — American University
Locations (1):
- American University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No